CLINICAL TRIAL: NCT03461003
Title: A Randomized Clinical Trial of the N-of-1 Approach in Children With Hypertension
Brief Title: N-of-1 Trials In Children With Hypertension
Acronym: NICHE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Joyce Philip Samuel, Assistant Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-17-1014; UL1TR003167 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-03-09 (Actual); Results first posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Hypertension
MeSH Terms: interventions — Amlodipine; Lisinopril; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NICHE method (Experimental): In the NICHE method, antihypertensive therapy will be chosen using an n-of-1 trial to identify the preferred therapy. Preferred therapy is defined a priori as that which produces the greatest reduction in ambulatory BP without intolerable side effects. Tested drugs will include amlodipine or losartan, lisinopril, and hydrochlorothiazide.
  Interventions: Other: NICHE method; Drug: Amlodipine; Drug: Lisinopril; Drug: Hydrochlorothiazide; Drug: Losartan
- Usual Care (Active Comparator): No protocol will be introduced to standardize BP management in the control arm.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: NICHE method — Based on underlying comorbidities at enrollment, patients will be assigned to either an unrestricted protocol (amlodipine versus lisinopril) or a restricted protocol (losartan versus lisinopril). Two drugs are tested in randomized order. Failure to achieve BP control at maximum doses of the first two drugs will result in augmentation with a diuretic (hydrochlorothiazide). BP control is assessed with 24 hour ambulatory monitoring at the end of each 2 week treatment period. Side effect tolerability is assessed with a questionnaire.
  Arms: NICHE method
Other: Usual care — Physician preference will dictate choice and adjustment of antihypertensive medication, BP measurement modality, interval between visits, and assessment of side effects.
  Arms: Usual Care
Drug: Amlodipine — Calcium-channel blocker; antihypertensive
  Arms: NICHE method
Drug: Lisinopril — Angiotensin-converting-enzyme (ACE) inhibitor; antihypertensive
  Arms: NICHE method
Drug: Hydrochlorothiazide — Thiazide diuretic; antihypertensive
  Arms: NICHE method
Drug: Losartan — Angiotensin II receptor blocker (ARB); antihypertensive
  Arms: NICHE method

SUMMARY:
The single patient (n-of-1) randomized trial is an underused approach to resolving therapeutic uncertainty by using a patient's own data to inform an individualized treatment plan. The proposed research is designed to assess whether the n-of-1 trial approach improves blood pressure control compared to usual care. This trial aims to advance learning about not only the treatment of pediatric hypertension but also the use of a neglected type of randomized trial to optimize the care of each patient.

DETAILED DESCRIPTION:
Pediatric hypertension, a growing problem, often requires prescription of antihypertensive medication. Pediatric hypertension specialists lack an evidentiary base on which to establish definitive clinical practice guidelines for first-line therapy. Significant practice variation is an unsurprising consequence. Routine choice of the same first-line therapy for most patients with hypertension, absent testing other options, may delay correction of blood pressure for months or years. Failure to incorporate patient preferences in medical decision-making may also contribute to decreased patient satisfaction and adherence.

Large parallel-group, comparative effectiveness trials are likely not on the horizon for this population. Moreover, heterogeneity of treatment effects would minimize the generalizability of such a trial to all patients.

This is a parallel-group, randomized clinical trial to compare the n-of-1 trial approach to usual care in normalizing blood pressure while minimizing exposure to compliance-reducing side effects.

ELIGIBILITY:
Inclusion Criteria:

* treating physician determines that pharmacologic therapy is indicated for treatment of hypertension
* ambulatory hypertension has been confirmed (off meds) within 12 months of enrollment

Exclusion Criteria:

* age < 10 years
* resistant hypertension (requiring ≥ 3 drug therapy)
* absolute contraindication or allergy to any of the tested drugs.

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2021-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce P. Samuel, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Derived] Samuel JP, Bell CS, Samuels JA, Rajan C, Walton AK, Green C, Tyson JE. N-of-1 Trials vs. Usual Care in Children With Hypertension: A Pilot Randomized Clinical Trial. Am J Hypertens. 2023 Feb 13;36(2):126-132. doi: 10.1093/ajh/hpac117. PMID 36227203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NICHE Method | Usual Care
Started | 23 | 26
Received Intervention | 21 | 22
Completed 6-month Follow up | 18 | 23
Completed | 18 | 23
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NICHE Method | Usual Care | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.9 [14.7 to 16.9] | 15.9 [14.4 to 16.8] | 15.9 [14.7 to 16.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 14 | 19 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic (black or white) | 17 | 18 | 35
  White (non-Hispanic) | 1 | 1 | 2
  Black (non-Hispanic) | 5 | 6 | 11
  Asian | 0 | 0 | 0
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49
Primary language of parent [Count of Participants; unit: Participants]
  English | 11 | 13 | 24
  Spanish | 12 | 13 | 25
Clinic Site [Count of Participants; unit: Participants]
  Multidisciplinary HTN clinic | 12 | 14 | 26
  County based clinic | 11 | 12 | 23
Hypertension type [Count of Participants; unit: Participants]
  Primary | 17 | 22 | 39
  Secondary | 6 | 4 | 10
Mean 24-hour ambulatory blood pressure at baseline (without medication) [Median (Inter-Quartile Range); unit: mm Hg] — To assess 24-hour ambulatory blood pressure, participants wear a 24-hour blood pressure monitor, which records blood pressure at regular intervals throughout a 24-hour period, while awake and while asleep. The mean of all recordings over the 24-hour period is calculated per participant, and the median of these means is reported. Population: Data not collected from 1 participant in the NICHE arm and 2 participants in the usual care arm
  mm Hg
    Systolic blood pressure: number analyzed (Participants) | 22 | 24 | 46
    Systolic blood pressure | 130 [126 to 133] | 130 [127 to 134] | 130 [127 to 134]
    Diastolic blood pressure: number analyzed (Participants) | 22 | 24 | 46
    Diastolic blood pressure | 76 [71 to 80] | 76 [74 to 81] | 76 [71 to 81]
BMI percentile for gender and age [Median (Full Range); unit: percentile] | 96.8 [10.5 to 99.8] | 95.8 [49.0 to 99.8] | 96 [10.5 to 99.8]
BMI categories [Count of Participants; unit: Participants]
  Underweight | 0 | 0 | 0
  Health weight | 4 | 6 | 10
  Overweight | 6 | 6 | 12
  Obese | 13 | 14 | 27
Number of participants with Chronic Kidney Disease [Count of Participants; unit: Participants] | 5 | 3 | 8
Number of participants with Diabetes Mellitus [Count of Participants; unit: Participants] | 2 | 2 | 4
Number of participants with Proteinuria [Count of Participants; unit: Participants] | 2 | 3 | 5
Number of participants who avoid calcium channel blocker [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ambulatory Blood Pressure (BP) Control at 6 Months
Description: Blood pressure control is when ambulatory blood pressure is normal, with normal as defined by the American Heart Association (AHA) criteria [the AHA criteria are systolic blood pressure and diastolic blood pressure (throughout wake and sleep) less than the 95th percentile based on the patient's gender and height]. To assess ambulatory blood pressure, participants wear a 24-hour blood pressure monitor, which records blood pressure at regular intervals throughout a 24-hour period.
Time Frame: 6 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 18 | 23
Participants
  Controlled | 8 | 8
  Uncontrolled | 10 | 15

2. Secondary Outcome: Change in Mean 24-hour Ambulatory Systolic Blood Pressure
Description: To assess 24-hour mean ambulatory blood pressure, participants wear a 24-hour blood pressure monitor, which records blood pressure at regular intervals throughout a 24-hour period, while awake and while asleep. The mean of all recordings over the 24-hour period is calculated per participant for both baseline and 6 months, and then the mean 24-hour systolic blood pressure at 6 months minus the mean 24-hour systolic blood pressure at baseline is calculated per participant. The average difference is reported, with a negative value indicating a reduction in blood pressure over time.
Time Frame: baseline, 6 months
Population: One patient in each arm was missing a baseline ambulatory blood pressure monitoring (ABPM), so change from baseline could not be calculated for each of those participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 17 | 22
mmHg | -10.6 (9.301) | -5.1 (9.586)

3. Secondary Outcome: Change in Mean Wake Ambulatory Systolic Blood Pressure
Description: To assess mean wake ambulatory blood pressure, participants wear a 24-hour blood pressure monitor, which records blood pressure at regular intervals throughout a 24 hour period, throughout wake and sleep. The mean of all recordings that occur while the participant is awake during the 24-hour period is calculated for both baseline and 6 months, and then the mean wake systolic blood pressure at 6 months minus the mean wake systolic blood pressure at baseline is calculated per participant. The average difference is reported, with a negative value indicating a reduction in blood pressure over time.
Time Frame: baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 17 | 22
mmHg | -10.5 (7.747) | -6.2 (10.123)

4. Secondary Outcome: Number of Participants Who Reported That Side Effects From Medication Led Them to Discontinue Medication
Time Frame: from baseline to 6 months
Population: Data were not collected from 5 participants in the NICHE method arm, and data were not collected from 5 participants in the Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 13 | 18
Participants | 0 | 3

5. Secondary Outcome: Number of Participants Who Self-reported Adherence to Intervention
Description: Adherence is reported as the number of participants who self-reported at the 6-month visit that they had not missed any doses of their medication in the preceding month.
Time Frame: from month 5 to month 6
Population: Data were not collected for 3 participants in the NICHE method arm.
Measure: Count of Participants; unit: Participants
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 15 | 23
Participants | 5 | 6

6. Secondary Outcome: Patient Satisfaction With Intervention as Assessed by a Survey
Description: Patient satisfaction is scored from 0 to 10, where 0 is the worst health care possible and 10 is the best health care possible.
Time Frame: 6 months
Population: Data were not collected for 4 participants in the NICHE method arm. Data were not collected for 2 participants in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NICHE Method | Usual Care
Number analyzed (Participants) | 14 | 21
score on a scale | 9.929 (0.267) | 9.667 (0.730)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | NICHE Method | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NICHE Method (N=23) | Usual Care (N=26)
Dizziness (Gastrointestinal disorders) | 0 | 1
Tiredness (General disorders) | 0 | 1
Sleeping Poorly (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03461003/Prot_SAP_002.pdf